CLINICAL TRIAL: NCT04223336
Title: A Web-enabled Integrated Care Pathway (ICP) for Addressing Multiple Modifiable Risk Factors as a Part of Smoking Cessation Treatment in Primary Care Settings.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government); Medical Psychiatry Alliance (Other)
Responsible Party: Principal Investigator, Peter Selby, Director, Medical Education, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 119-2018
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Physical Activity; Fruits and Vegetable Consumption; Smoking Cessation
Keywords: smoking cessation; physical activity; diet; primary care; screening; brief intervention; integrated care pathway
MeSH Terms: conditions — Motor Activity; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Individuals enrolling into the STOP program at a primary care organization (Family Health Team, Community Health Centre, or Nurse Practitioner-led Clinic) will be randomly allocated in a 1:1 allocation ratio to control or intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): When a participant in the control group is identified via a mandatory baseline questionnaire as having low levels of physical activity and/or low levels of fruits/vegetable consumption, the practitioner seeing this participant during their visit will not receive any computer alerts for physical activity and fruits/vegetable consumption. However, practitioners will still have access to the physical activity and diet data as part of the baseline assessment (Screening). Practitioners will also continue to have access to all the same resources as they currently do (treatment as usual).
- Intervention Group (Experimental): When a participant in the intervention group is identified via mandatory baseline questionnaire as having low levels of physical activity and/or low levels of fruits/vegetable consumption, the practitioner seeing this participant during their visit will receive computer alerts (screening), prompting to provide participant with a brief intervention (risk communication) and a self-monitoring resource for physical activity and/or fruits/vegetable consumption.
  Interventions: Behavioral: Brief physical activity and diet intervention

INTERVENTIONS:
Behavioral: Brief physical activity and diet intervention — The intervention is an integrated care pathway that provides a computerized prompts for practitioners in the STOP program via their online portal. For a participant who is in the intervention group, the online portal will screen the participant for their physical activity and fruit/vegetable consumption and provide the practitioner (who is seeing this participant for their visit) with computerized alerts for physical activity and fruits/vegetable consumption. Specifically, the portal will prompt practitioners to provide a brief intervention for these two behaviours using risk communication and will also suggest brief intervention language designed based on the Elicit-Provide-Elicit framework. The portal will also have available a self-monitoring resource for physical activity and fruits/vegetable consumption and will prompt practitioners to provide this self-monitoring resource to the participant during their visit.
  Arms: Intervention Group

SUMMARY:
Compared to non-smokers, smokers are significantly more likely to also engage in other chronic disease-related risk behaviours; which can be a barrier to quitting successfully. Therefore a holistic approach is needed for smoking cessation treatment. The Smoking Treatment for Ontario Patients (STOP) program currently offers an online integrated care pathway (ICP) for addressing alcohol and mood as a part of smoking cessation treatment. Evidence also shows that smokers are also more likely to be physical inactive and not consume enough fruits/vegetables. These risk behaviours can further compound the negative health effects for smokers. However, it is remains unclear which and how many behaviours should be addressed simultaneously in smoking cessation treatment and what the impact on smoking cessation and care for STOP participants will be.

Through this study, the investigators will seek to:

1. Determine whether the addition of an integrated care pathway for physical activity and fruits/vegetable consumption to the STOP program is associated with participants' quit prevalence at 6 month follow-up among STOP participants who are physically inactive and/or have low levels of fruits/vegetable consumption.
2. Understand how the integrated care pathway for physical activity and fruits/vegetable consumption is implemented in primary care settings. In the process, we hope to generate insights on how this ICP can be most helpful to organizations, staff and patients.

DETAILED DESCRIPTION:
Tobacco use, in particular, continues to be the leading cause of preventable death, with a recent review identifying strong associations between tobacco and other modifiable risk behaviours. Tobacco users tend to consume more alcohol, eat less fruits and vegetables and report less minutes of leisure physical activity as compared with non-tobacco users. The clustering of these modifiable risk behaviours among tobacco users not only translates a heightened risk for cardiovascular disease but may also negatively influence the likelihood of successful smoking cessation. Alcohol consumed even in small amounts, has been shown to increase cravings for smoking, thus increasing risk of relapse to smoking. Increasing physical activity levels can help to reduce tobacco withdrawal and cravings, as well as minimize the reward anticipation. Individuals also often misattribute the reversal of withdrawal symptoms (i.e. irritability) from smoking as relief from stress. This can also increase the risk of relapse when attempting to quit.

In addition to the more direct relationships between these health behaviours and smoking cessation, successfully changing one or more behaviours may also help to increase self-efficacy and self-confidence to change other health behaviours that individuals may be less motivated to act on. As a result, targeting multiple risk behaviours in smokers may help maximize health promotion efforts by augmenting smoking abstinence rates, improving overall health, and reducing healthcare-related costs. In order to address this, the Smoking Treatment for Ontario Patients (STOP) Program (REB#: 058-2011), a province-wide initiative that uses the existing healthcare infrastructure to provide smoking cessation support to smokers in Ontario, has been developed and is currently testing a web-enabled Integrated Care Pathways (ICP) for some of these behaviours. In 2016, the STOP program started offering specialized clinical pathways through the STOP Portal (a web-based platform and an online data collection/management tool used by the STOP practitioners to complete participant enrollment and record smoking status at each visit) for smokers who drink above Canadian Cancer Society guidelines (REB# 035-2015). In 2018, it added a specialized ICP for those who have mood disorders (REB#: 065-2016). However, there are currently no web-enabled tools in the STOP program that also address some of the other well-known modifiable risk factors such as: physical activity, and diet.

There is substantial high quality evidence that shows the effectiveness of screening for these behaviors, providing a brief intervention, and referral to treatment when needed for helping patients quit smoking as well as change other behaviours. Moreover, a recent systematic review of behaviour change techniques practitioners can use to promote health behaviour change in patients found that, relative to other techniques, 'risk communication' and 'self-monitoring of behaviour' are the most effective techniques.

As a result, we designed the intervention - an integrated care pathway that facilitates practitioners to deliver a brief intervention that includes risk communication, and provides tools for patients to monitor their health behaviours to STOP patients who have at least one of the following other modifiable risk factors at baseline: low levels of physical activity, and low levels of fruits/vegetable consumption. Low levels of physical activity will be defined as being below the Canadian national guidelines: less than 150 min per week of moderate-to-vigorous activity. Low fruits and vegetable is defined as being below the 2007 Canada's Food Guide: less than 7 servings (female) or 8 servings (male) of fruits/vegetable per day.

The specific components of the intervention are outlined below:

1. Systematic screening through the STOP portal for STOP participants with at least one of the following risk factors: low levels of physical activity, and low fruits/vegetable consumption.
2. Have computer prompts that advise the practitioner of patient's risk factors, and to provide a brief intervention that includes how the identified risk factors affect the patient's ability to quit successfully (Risk communication).
3. Provision of self-monitoring tool(s) for monitoring physical activity and/or fruits/vegetable consumption levels.

This study aims to assess whether the addition of an ICP for physical activity and diet into Family Health Teams (FHTs), Community Health Centres (CHCs), and Nurse Practitioner-led Clinics (NPLCs) participating in the STOP program is associated with participants' quit rate at 6 month follow-up. Individuals enrolling into the STOP program through one of these organizations will be randomly allocated (1:1) to control vs intervention group. In addition, we hope to gather insights on how this ICP can be most helpful to organizations, staff and patients, thereby informing implementation processes in other primary care settings across Canada/ Ontario. Our evaluation includes patient, clinician, and organization-level outcomes. To organize this multifaceted evaluation, we use the Reach, Efficacy, Adoption, Implementation, and Maintenance (RE-AIM) framework.

ELIGIBILITY:
Inclusion Criteria:

The sample of patients for the study will be recruited from 153 Family Health Teams (FHTs), 61 Community Health Centres (CHCs) and 18 Nurse Practitioner-Led Clinics (NPLCs) currently participating in the STOP program. The inclusion criteria are as follows:

* An individual enrolling in the STOP program at a participating FHT, CHC, or NPLC.
* Must have at least one of the following two modifiable risk factors: low levels of physical activity and/or low levels of fruits/vegetable consumption.
* Enrollment into STOP program must be completed online on the STOP Portal, in real-time with the participant present.
* Must have at least one piece of contact information (e.g. phone number or email address).

Exclusion Criteria:

* An individual enrolling in the STOP program at a participating Addictions Agencies (AAs)
* STOP enrollment conducted on paper, no contact information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5331 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2021-05-02 (Actual); Study Completion 2021-05-02 (Actual)

PRIMARY OUTCOMES:
Smoking cessation - self-report questionnaire | 6-month follow-up
  The primary outcome of the study, measured at the patient level, is 7 day point prevalence of abstinence at 6 month follow-up. We will compare the proportion of intervention vs control group participants who report being quit at follow-up.

SECONDARY OUTCOMES:
Physical activity - self-report questionnaire | 6-month follow-up
  The secondary outcome, also measured at the patient level, is change in physical activity levels from baseline to 6 months follow-up. We will compare the change in physical activity from baseline to 6 month follow-up in intervention vs control group participants.
Fruits/vegetable consumption - self-report questionnaire | 6-month follow-up
  The secondary outcome, also measured at the patient level, is change in fruits/vegetable consumption levels from baseline to 6 months follow-up. We will compare the change in fruits/vegetable consumption levels from baseline to 6 month follow-up in intervention vs control group participants.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Selby, MBBS CCFP FCFP MHSc DipABAM, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Minian N, Mehra K, Lingam M, Dragonetti R, Veldhuizen S, Zawertailo L, deRuiter WK, Melamed OC, Moineddin R, Thorpe KE, Taylor VH, Hahn M, Selby P. Healthcare providers' perspectives on implementing a brief physical activity and diet intervention within a primary care smoking cessation program: a qualitative study. BMC Prim Care. 2024 Jan 6;25(1):16. doi: 10.1186/s12875-023-02259-3. PMID 38184559
- [Derived] Minian N, Lingam M, Moineddin R, Thorpe KE, Veldhuizen S, Dragonetti R, Zawertailo L, Taylor VH, Hahn M, deRuiter WK, Melamed OC, Selby P. The Impact of a Clinical Decision Support System for Addressing Physical Activity and Healthy Eating During Smoking Cessation Treatment: Hybrid Type I Randomized Controlled Trial. J Med Internet Res. 2022 Sep 30;24(9):e37900. doi: 10.2196/37900. PMID 36178716
- [Derived] Minian N, Lingam M, Moineddin R, Thorpe KE, Veldhuizen S, Dragonetti R, Zawertailo L, Taylor VH, Hahn M, deRuiter WK, Melamed O, Selby P. Impact of a Web-Based Clinical Decision Support System to Assist Practitioners in Addressing Physical Activity and/or Healthy Eating for Smoking Cessation Treatment: Protocol for a Hybrid Type I Randomized Controlled Trial. JMIR Res Protoc. 2020 Sep 29;9(9):e19157. doi: 10.2196/19157. PMID 32990250